CLINICAL TRIAL: NCT01767987
Title: Ranolazine Cardioprotection in PCI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study due to lack of enrollment
Sponsor: Harvey Hahn (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Harvey Hahn, Director, Cardiovascular Fellowship Training Program and Director, Cardiac Noninvasive Laboratory, Kettering Health Network
Organization: Kettering Health Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ISR IN-US-259-0139
Record Dates: First submitted 2012-11-28; First posted 2013-01-15 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; ACS; Percutaneous Coronary Intervention; PCI; Ranolazine; Coronary Angiogram; Cardioprotectant
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): Oral treatment Intervention: Drug: Ranolazine 1000 mg
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Oral treatment Intervention: Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Drug: Ranolazine 1000 mg Oral dose twice per day for 3 days leading up to PCI
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Drug: Placebo Oral dose twice per day for 3 days leading up to PCI
  Arms: Placebo

SUMMARY:
The investigators will test if upfront dosing of Ranolazine can reduce myocardial biomarker release (CK-MB, Troponin) post percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Ranolazine has been demonstrated to decrease angina, ischemia on perfusion imaging, improve diastolic function, and cardiac metabolism. Furthermore it has been associated with reduced cardiac arrhythmias, including non-sustained ventricular tachycardia and atrial fibrillation. It has not been studied as an acute cardioprotective agent in percutaneous coronary intervention (PCI).

We hypothesize that upfront administration of Ranolazine could decrease the myocardial injury associated with PCI due to all the factors listed above (i.e. precondition the myocardium). We plan to screen all patients scheduled for an elective coronary angiogram. Those who meet criteria and consent will be randomized to either receive Ranolazine or placebo twice a day for 3 days leading up to the PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients undergoing Coronary Angiography with possible PCI
* Able and willing to give consent
* Able to read and write English

Exclusion Criteria:

* Current EKG or Biomarker of Acute Myocardial Infarction (MI) or Acute Coronary Syndromes (ACS)
* History of Allergy to Ranolazine
* Pregnant or Nursing
* Currently taking Ranolazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Hahn, MD, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 4 | 2
Completed | 0 | 1
Not Completed | 4 | 1
Not completed — Physician Decision | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [51 to 66] | 67.5 [65 to 70] | 63.5 [51 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Troponin
Description: Troponin labs will be drawn 8-10 hrs after PCI or at discharge whichever comes first
Time Frame: 8-10 hrs post PCI
Population: Of the 4 Ranolazine Group subjects, 1 was withdrawn for pre-procedure study drug non-compliance; 3 had no PCI intervention. Of the 2 Placebo Group subject, 1 had no PCI intervention. The only subject undergoing PCI intervention was from the Placebo Group and was thus the only subject undergoing this protocol required test.
Measure: Number; unit: NG/ML
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
NG/ML |  | 0.023

2. Primary Outcome: CK-MB
Description: CK-MB labs will be drawn 8-10 hrs after PCI or at discharge whichever comes first
Time Frame: 8-10 hrs post PCI
Population: For the single subject completing the PCI intervention, CK-MB was not done because the CK level was below the threshold running the CK-MB test.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: TIMI Flow Rate (Grade)
Description: This TIMI classification was developed by the TIMI (Thrombolysis In Myocardial Infarction) study group to semiquantitatively assess coronary artery perfusion beyond point of occlusion on coronary angiography.* TIMI Grade [Description] TIMI 0 - no perfusion [no antegrade flow beyond the point of occlusion] TIMI 1 - penetration without perfusion [faint antegrade coronary flow beyond the occlusion with incomplete filling of the distal coronary bed] TIMI 2 - partial perfusion [delayed or sluggish antegrade flow with complete filling of the distal territory] TIMI 3 - complete perfusion [normal flow with complete filling of the distal territory]
  *(see http://radclass.mudr.org/content/timi-grade-flow-grading-coronary-blood-flow-during-coronary-angiography) TIMI 0 is the least favorable grade. TIMI 3 is the most favorable grade.
Time Frame: TIMI Flow Rate (Grade) is assessed immediately after an interventional reperfusion attempt during a PCI (Percutaneous Coronary Intervention) procedure.
Population: The only subject undergoing PCI intervention was from the Placebo Group and was thus the only subject for whom this protocol required data point was collected.
Measure: Number; unit: units on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
units on a scale |  | 3

4. Secondary Outcome: Incidence of Atrial Fibrillation, Ventricular Tachycardia, or Ventricular Fibrillation in Coronary Cath Lab
Description: Abnormal heart activity
Time Frame: During the PCI (Percutaneous Coronary Intervention) procedure - starting at timepoint of guidewire insertion into the access artery until removal of guidewire
Population: The only subject undergoing PCI intervention was from the Placebo Group and was thus the only subject for whom these protocol required data points were collected.
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
participants |  | 0

5. Secondary Outcome: Incidence of Non-sustained Ventricular Tachycardia or Atrial Fibrillation Post PCI
Time Frame: Following completion of PCI through hospital discharge
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
participants |  | 0

6. Secondary Outcome: Left Ventricular End Diastolic Pressure (LVEDP)
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Number; unit: mmHG
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
mmHG |  | 10

7. Secondary Outcome: Death, Myocardial Infarction (Biomarker Greater Than 2x Normal), CHF, Cardiac Arrest
Time Frame: At discharge or within 1 days, whichever comes first
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
participants |  | 0

8. Secondary Outcome: Death, MI, Revascularization, CHF
Time Frame: 1-4 weeks post PCI
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
participants |  | 0

9. Secondary Outcome: Successful PCI
Description: For the purposes of this study, a successful PCI is considered one where no additional coronary interventions were required within 24 hours after the initial PCI.
Time Frame: At discharge or within 1 days, whichever comes first
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 1
participants |  | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of consent through end of study discharge from hospital. Adverse events unresolved at discharge were to be followed to resolution. No events occuring after discharge were to be recorded as adverse events.
Description: Study timeline consisted of consent, pre-procedure medication (3 days), arrival for out-patient heart cath procedure, possible PCI, post-procedure recovery time, and discharge from hospital recovery room. Time from consent to start of study meds varied. Time from start of study drug to discharge was 4 days.
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes